CLINICAL TRIAL: NCT05285969
Title: Motivational Interview for Cardiac Rehabilitation in Acute Myocardial Infarction: A Randomized Controlled Trial in the Primary Healthcare Area.
Brief Title: Cardiac Rehabilitation With Motivational Interview for Acute Myocardial Infarction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Consorci d'Atenció Primària de Salut de l'Eixample (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Institut Català de la Salut (Other); Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other); Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other); Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Luis Gonzalez de Paz, Researcher, Consorci d'Atenció Primària de Salut de l'Eixample
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCB/2019/0727
Record Dates: First submitted 2022-02-28; First posted 2022-03-18 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Myocardial Infarction, Acute
Keywords: Myocardial Infarction; Cardiac Rehabilitation; Rehabilitation Nursing; Primary Health Care; Motivational Interviewing
MeSH Terms: conditions — Myocardial Infarction | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational interview (Experimental): Motivation Interview program with standard care
  Interventions: Behavioral: Motivational interview
- Standard care group (Active Comparator): Standard care
  Interventions: Behavioral: Active Comparator: Standard care group

INTERVENTIONS:
Behavioral: Motivational interview — The new CR program with MI will be structured in 4 sessions and an optional fifth during the six months after discharge. The methodology of the MI sessions will follow the four phases logical sequence of MI proposed by Rollnick and Millner. 1) engage in a collaborative relationship, 2) focus on a particular change, 3) evoke intrinsic motivations for change, and 4) plan an immediate step for change
  Arms: Motivational interview
Behavioral: Active Comparator: Standard care group — All patients in the control group will receive a kit with informative material with the actions and procedures to follow (diet, physical activity, smoking cessation, and other recommendations about secondary prevention).
  Arms: Standard care group

SUMMARY:
Introduction: Secondary prevention after acute myocardial infarction may include cardiac rehabilitation and lifestyle changes. Cardiac rehabilitation has mainly taken place in hospitals without coordination with primary healthcare. Motivational interviews have been shown to be effective as a means for change in patients after acute myocardial infarction. The objective of this study is to evaluate the effectiveness of a cardiac rehabilitation program with motivational interviews in patients discharged from hospital after acute myocardial infarction.

Methods: Randomized clinical non-pharmacological trial. A minimum sample of 284 participants requiring cardiac rehabilitation after acute myocardial infarction in six primary healthcare centers. Participants will be randomized to cardiac rehabilitation with motivational interviews or normal standard of care. All secondary results will be evaluated at 1,3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Hospital admission for acute coronary syndrome (diagnostic codes ICD-10: I20-I22).
* Post unscheduled cardiac revascularization surgery (procedure code ICD-10: 021x).
* Discharge to home with the area of the 7 PHCs.
* Indication of RC indication.
* Voluntary participation.

Exclusion Criteria:

* Acute aortic disease,
* Severe pulmonary hypertension.
* Uncontrolled arrhythmias.
* Decompensated Heart Failure or significant valvular or congenital heart disease.
* Intervention in heart valves and/or interventricular septum.
* Diseases that prevent exercise.
* Osteoarticular disease that severely limits exercise.
* Severe mental disorder.
* Any severe psychiatric disorders.
* Cognitive disability.
* Verbal communication problems.
* Participation in hospital Cardiac Rehabilitation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Physical functional capacity | 1st month
  Improvement in aerobic capacity and resistance, measured by a physical effort test
Physical functional capacity | 6th month
  Improvement in aerobic capacity and resistance, measured by a physical effort test

SECONDARY OUTCOMES:
Effectiveness of secondary prevention | 1st month
  Effectiveness of secondary prevention will be considered (Satisfied / no satisfied) with next conditions (all together):
  Blood pressure values <140/90mmHg, plasma cholesterol c-LDL<70mg/dL, plasma glycosylated hemoglobin <7%. Absolute cessation or no initiation of smoking Body Mass Index in the range of 18.5-25kg/m^2.
Effectiveness of secondary prevention | 3rd month
  Effectiveness of secondary prevention will be considered (Satisfied / no satisfied) with next conditions (all together):
  Blood pressure values <140/90mmHg, plasma cholesterol c-LDL<70mg/dL, plasma glycosylated hemoglobin <7%. Absolute cessation or no initiation of smoking Body Mass Index in the range of 18.5-25kg/m^2.
Effectiveness of secondary prevention | 6th month
  Effectiveness of secondary prevention will be considered (Satisfied / no satisfied) with next conditions (all together):
  Blood pressure values <140/90mmHg, plasma cholesterol c-LDL<70mg/dL, plasma glycosylated hemoglobin <7%. Absolute cessation or no initiation of smoking Body Mass Index in the range of 18.5-25kg/m^2.
Psychological status | 6th month
  Measured with the Psychological General Well-Being Index (PGWBI)
Perceived quality of life | 1st month
  Physical and mental summaries of perceived quality of life measured with the generic quality of life Short Form questionnaire (SF-12).
Perceived quality of life | 2nd month
  Physical and mental summaries of perceived quality of life measured with the generic quality of life Short Form questionnaire (SF-12).
Perceived quality of life | 3rd month
  Physical and mental summaries of perceived quality of life measured with the generic quality of life Short Form questionnaire (SF-12).

CONTACTS AND LOCATIONS:
Overall Officials: Luis González de Paz, PhD, Principal Investigator — Consorci d'Atenció Primària de Salut Barcelona Esquerra (CAPSBE); Rocío Rodríguez Romero, RN, Study Chair — Consorci d'Atenció Primària de Salut Barcelona Esquerra (CAPSBE); Carles Falces Salvador, PhD, Study Chair — Cardiovascular Institute. Hospital Clínic. University of Barcelona, Barcelona, Spain.
Locations (4):
- Spain (4):
  - Centre Atenció Primària de Les Corts, Barcelona
  - CAP Compte Borrell, Barcelona
  - Centre Atenció Primària Montengre, Barcelona
  - Centre Atenció Primària Casanova, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bjarnason-Wehrens B, McGee H, Zwisler AD, Piepoli MF, Benzer W, Schmid JP, Dendale P, Pogosova NG, Zdrenghea D, Niebauer J, Mendes M; Cardiac Rehabilitation Section European Association of Cardiovascular Prevention and Rehabilitation. Cardiac rehabilitation in Europe: results from the European Cardiac Rehabilitation Inventory Survey. Eur J Cardiovasc Prev Rehabil. 2010 Aug;17(4):410-8. doi: 10.1097/HJR.0b013e328334f42d. PMID 20300001
- [Background] Abreu A, Pesah E, Supervia M, Turk-Adawi K, Bjarnason-Wehrens B, Lopez-Jimenez F, Ambrosetti M, Andersen K, Giga V, Vulic D, Vataman E, Gaita D, Cliff J, Kouidi E, Yagci I, Simon A, Hautala A, Tamuleviciute-Prasciene E, Kemps H, Eysymontt Z, Farsky S, Hayward J, Prescott E, Dawkes S, Pavy B, Kiessling A, Sovova E, Grace SL. Cardiac rehabilitation availability and delivery in Europe: How does it differ by region and compare with other high-income countries?: Endorsed by the European Association of Preventive Cardiology. Eur J Prev Cardiol. 2019 Jul;26(11):1131-1146. doi: 10.1177/2047487319827453. Epub 2019 Feb 20. PMID 30782007
- [Background] Martín R. Efectividad de la rehabilitación cardíaca en un grupo de pacientes de alto riesgo. Rev Enferm Cardiol. 2018;25(75):34-39.
- [Background] Shields GE, Wells A, Doherty P, Heagerty A, Buck D, Davies LM. Cost-effectiveness of cardiac rehabilitation: a systematic review. Heart. 2018 Sep;104(17):1403-1410. doi: 10.1136/heartjnl-2017-312809. Epub 2018 Apr 13. PMID 29654096
- [Background] Piepoli MF, Corra U, Adamopoulos S, Benzer W, Bjarnason-Wehrens B, Cupples M, Dendale P, Doherty P, Gaita D, Hofer S, McGee H, Mendes M, Niebauer J, Pogosova N, Garcia-Porrero E, Rauch B, Schmid JP, Giannuzzi P. Secondary prevention in the clinical management of patients with cardiovascular diseases. Core components, standards and outcome measures for referral and delivery: a policy statement from the cardiac rehabilitation section of the European Association for Cardiovascular Prevention & Rehabilitation. Endorsed by the Committee for Practice Guidelines of the European Society of Cardiology. Eur J Prev Cardiol. 2014 Jun;21(6):664-81. doi: 10.1177/2047487312449597. Epub 2012 Jun 20. PMID 22718797
- [Background] Verbo E. Protocolo de rehabilitación cardiaca en pacientes con insuficiencia cardiaca (Tesis). Universidad CEU-San Pablo. 2012.
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Background] Kotseva K, Wood D, De Bacquer D, De Backer G, Ryden L, Jennings C, Gyberg V, Amouyel P, Bruthans J, Castro Conde A, Cifkova R, Deckers JW, De Sutter J, Dilic M, Dolzhenko M, Erglis A, Fras Z, Gaita D, Gotcheva N, Goudevenos J, Heuschmann P, Laucevicius A, Lehto S, Lovic D, Milicic D, Moore D, Nicolaides E, Oganov R, Pajak A, Pogosova N, Reiner Z, Stagmo M, Stork S, Tokgozoglu L, Vulic D; EUROASPIRE Investigators. EUROASPIRE IV: A European Society of Cardiology survey on the lifestyle, risk factor and therapeutic management of coronary patients from 24 European countries. Eur J Prev Cardiol. 2016 Apr;23(6):636-48. doi: 10.1177/2047487315569401. Epub 2015 Feb 16. PMID 25687109
- [Background] Haykowsky M, Scott J, Esch B, Schopflocher D, Myers J, Paterson I, Warburton D, Jones L, Clark AM. A meta-analysis of the effects of exercise training on left ventricular remodeling following myocardial infarction: start early and go longer for greatest exercise benefits on remodeling. Trials. 2011 Apr 4;12:92. doi: 10.1186/1745-6215-12-92. PMID 21463531
- [Background] Bohplian S, Bronas UG. Motivational Strategies and Concepts to Increase Participation and Adherence in Cardiac Rehabilitation: AN INTEGRATIVE REVIEW. J Cardiopulm Rehabil Prev. 2022 Mar 1;42(2):75-83. doi: 10.1097/HCR.0000000000000639. PMID 34753873
- [Background] Sociedad Española de Cardiología. Registro Nacional de Unidades de Rehabilitación Cardíaca. R- EUReCa. Available from: https://secardiologia.es/riesgo/cientifico/6415-registro-nacional-de-unidades-de-rehabilitacion- cardiaca-r-eureka (accessed 30 Jan 2019).
- [Background] Rodrigo-Banos V, Moral-Pairada MD, Gonzalez-de Paz L. A Comprehensive Assessment of Informal Caregivers of Patients in a Primary Healthcare Home-Care Program. Int J Environ Res Public Health. 2021 Nov 4;18(21):11588. doi: 10.3390/ijerph182111588. PMID 34770102
- [Background] Gene-Badia J, Ascaso C, Escaramis-Babiano G, Sampietro-Colom L, Catalan-Ramos A, Sans-Corrales M, Pujol-Ribera E. Personalised care, access, quality and team coordination are the main dimensions of family medicine output. Fam Pract. 2007 Feb;24(1):41-7. doi: 10.1093/fampra/cml056. Epub 2006 Nov 1. PMID 17079249
- [Background] Pujol Ribera E, Gene Badia J, Sans Corrales M, Sampietro-Colom L, Pasarin Rua MI, Iglesias-Perez B, Casajuana-Brunet J, Escaramis-Babiano G. [Primary health care product defined by health professionals and users]. Gac Sanit. 2006 May-Jun;20(3):209-19. doi: 10.1157/13088852. Spanish. PMID 16756859
- [Background] Palomo L, Gene-Badia J, Rodriguez-Sendin JJ. [The reform of primary care, between the last refuge of adventure and innovation. SESPAS report 2012]. Gac Sanit. 2012 Mar;26 Suppl 1:14-9. doi: 10.1016/j.gaceta.2011.06.010. Epub 2011 Oct 11. Spanish. PMID 21996448
- [Background] Santesmases-Masana R, Gonzalez-de Paz L, Hernandez-Martinez-Esparza E, Kostov B, Navarro-Rubio MD. Self-Care Practices of Primary Health Care Patients Diagnosed with Chronic Heart Failure: A Cross-Sectional Survey. Int J Environ Res Public Health. 2019 May 9;16(9):1625. doi: 10.3390/ijerph16091625. PMID 31075932
- [Background] Buckingham SA, Taylor RS, Jolly K, Zawada A, Dean SG, Cowie A, Norton RJ, Dalal HM. Home-based versus centre-based cardiac rehabilitation: abridged Cochrane systematic review and meta-analysis. Open Heart. 2016 Sep 14;3(2):e000463. doi: 10.1136/openhrt-2016-000463. eCollection 2016. PMID 27738516
- [Background] Poudel N, Kavookjian J, Scalese MJ. Motivational Interviewing as a Strategy to Impact Outcomes in Heart Failure Patients: A Systematic Review. Patient. 2020 Feb;13(1):43-55. doi: 10.1007/s40271-019-00387-6. PMID 31502239
- [Background] Taylor RS, Dalal H, Jolly K, Moxham T, Zawada A. Home-based versus centre-based cardiac rehabilitation. Cochrane Database Syst Rev. 2010 Jan 20;(1):CD007130. doi: 10.1002/14651858.CD007130.pub2. PMID 20091618
- [Background] Dalal HM, Doherty P, Taylor RS. Cardiac rehabilitation. BMJ. 2015 Sep 29;351:h5000. doi: 10.1136/bmj.h5000. No abstract available. PMID 26419744
- [Background] Arena R, Williams M, Forman DE, Cahalin LP, Coke L, Myers J, Hamm L, Kris-Etherton P, Humphrey R, Bittner V, Lavie CJ; American Heart Association Exercise, Cardiac Rehabilitation and Prevention Committee of the Council on Clinical Cardiology, Council on Epidemiology and Prevention, and Council on Nutrition, Physical Activity and Metabolism. Increasing referral and participation rates to outpatient cardiac rehabilitation: the valuable role of healthcare professionals in the inpatient and home health settings: a science advisory from the American Heart Association. Circulation. 2012 Mar 13;125(10):1321-9. doi: 10.1161/CIR.0b013e318246b1e5. Epub 2012 Jan 30. No abstract available. PMID 22291128
- [Background] Sakane K, Kanzaki Y, Ito T, Hoshiga M. Motivational interviewing as a new approach to improve outcome through self-care behavioural changes in advanced heart failure patient: a case report. Eur Heart J Case Rep. 2021 Oct 1;5(10):ytab395. doi: 10.1093/ehjcr/ytab395. eCollection 2021 Oct. PMID 34738065
- [Background] Jokar F, Yousefi H, Yousefy A, Sadeghi M. Begin Again and Continue With Life: A Qualitative Study on the Experiences of Cardiac Rehabilitation Patients. J Nurs Res. 2017 Oct;25(5):344-352. doi: 10.1097/JNR.0000000000000220. PMID 28877121
- [Background] Masterson Creber R, Patey M, Lee CS, Kuan A, Jurgens C, Riegel B. Motivational interviewing to improve self-care for patients with chronic heart failure: MITI-HF randomized controlled trial. Patient Educ Couns. 2016 Feb;99(2):256-64. doi: 10.1016/j.pec.2015.08.031. Epub 2015 Aug 29. PMID 26358533
- [Background] Hardcastle SJ, Taylor AH, Bailey MP, Harley RA, Hagger MS. Effectiveness of a motivational interviewing intervention on weight loss, physical activity and cardiovascular disease risk factors: a randomised controlled trial with a 12-month post-intervention follow-up. Int J Behav Nutr Phys Act. 2013 Mar 28;10:40. doi: 10.1186/1479-5868-10-40. PMID 23537492
- [Background] Wood DA, Kotseva K, Connolly S, Jennings C, Mead A, Jones J, Holden A, De Bacquer D, Collier T, De Backer G, Faergeman O; EUROACTION Study Group. Nurse-coordinated multidisciplinary, family-based cardiovascular disease prevention programme (EUROACTION) for patients with coronary heart disease and asymptomatic individuals at high risk of cardiovascular disease: a paired, cluster-randomised controlled trial. Lancet. 2008 Jun 14;371(9629):1999-2012. doi: 10.1016/S0140-6736(08)60868-5. PMID 18555911
- [Background] Paradis V, Cossette S, Frasure-Smith N, Heppell S, Guertin MC. The efficacy of a motivational nursing intervention based on the stages of change on self-care in heart failure patients. J Cardiovasc Nurs. 2010 Mar-Apr;25(2):130-41. doi: 10.1097/JCN.0b013e3181c52497. PMID 20168193
- [Background] Vellone E, Rebora P, Ausili D, Zeffiro V, Pucciarelli G, Caggianelli G, Masci S, Alvaro R, Riegel B. Motivational interviewing to improve self-care in heart failure patients (MOTIVATE-HF): a randomized controlled trial. ESC Heart Fail. 2020 Jun;7(3):1309-1318. doi: 10.1002/ehf2.12733. Epub 2020 Apr 28. PMID 32343483
- [Background] Flores PVP, Rocha PA, Figueiredo LDS, Guimaraes TML, Velasco NS, Cavalcanti ACD. Effect of motivational interviewing on self-care of people with heart failure: a randomized clinical trial. Rev Esc Enferm USP. 2020 Nov 6;54:e03634. doi: 10.1590/S1980-220X2019013703634. eCollection 2020. English, Portuguese. PMID 33175022
- [Background] Sokalski T, Hayden KA, Raffin Bouchal S, Singh P, King-Shier K. Motivational Interviewing and Self-care Practices in Adult Patients With Heart Failure: A Systematic Review and Narrative Synthesis. J Cardiovasc Nurs. 2020 Mar/Apr;35(2):107-115. doi: 10.1097/JCN.0000000000000627. PMID 31851149
- [Background] Chew HSJ, Cheng HY, Chair SY. The suitability of motivational interviewing versus cognitive behavioural interventions on improving self-care in patients with heart failure: A literature review and discussion paper. Appl Nurs Res. 2019 Feb;45:17-22. doi: 10.1016/j.apnr.2018.11.006. Epub 2018 Nov 7. PMID 30683246
- [Background] Brodie DA, Inoue A, Shaw DG. Motivational interviewing to change quality of life for people with chronic heart failure: a randomised controlled trial. Int J Nurs Stud. 2008 Apr;45(4):489-500. doi: 10.1016/j.ijnurstu.2006.11.009. Epub 2007 Jan 26. PMID 17258218
- [Derived] Rodriguez-Romero R, Falces C, Kostov B, Garcia-Planas N, Blat-Guimera E, Alvira-Balada MC, Lopez-Poyato M, Benito-Serrano ML, Vidiella-Pinol I, Zamora-Sanchez JJ, Benet M, Garnacho-Castano MV, Santos-Ruiz S, Santesmases-Masana R, Roura-Rovira S, Benavent-Areu J, Siso-Almirall A, Gonzalez-de Paz L. A motivational interview program for cardiac rehabilitation after acute myocardial infarction: study protocol of a randomized controlled trial in primary healthcare. BMC Prim Care. 2022 May 6;23(1):106. doi: 10.1186/s12875-022-01721-y. PMID 35513777